CLINICAL TRIAL: NCT00935792
Title: Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL) With Everolimus (RAD001) and Alemtuzumab: A Phase I/II Study
Brief Title: Everolimus and Alemtuzumab in Treating Patients With Recurrent Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC088C; MC088C (Other: Mayo Clinic Cancer Center); NCI-2009-00935 (Registry Identifier: NCI's CTRO); 08-008775 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-07-06; First posted 2009-07-09 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2016-01

CONDITIONS: Lymphocytic Leukemia
Keywords: hematopoietic cancer; lymphoid cancer
MeSH Terms: conditions — Leukemia, Lymphoid; Hematologic Neoplasms | interventions — Alemtuzumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 8 weeks.
  Interventions: Drug: alemtuzumab; Drug: everolimus

INTERVENTIONS:
Drug: alemtuzumab — Given subcutaneously
  Other Names: anti-CD52 monoclonal antibody; MoAb CD52; Monoclonal Antibody Campath-1H; Campath-1H; Monoclonal Antibody CD52; Campath
Drug: everolimus — Given orally
  Other Names: Certican; RAD001; 42-O-(2-Hydroxy)ethyl Rapamycin

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the signaling molecules needed for cell growth. Monoclonal antibodies, such as alemtuzumab, can bind to and kill malignant lymphocytes.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus when given together with alemtuzumab and will see how well they work in treating patients with recurrent chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Test the safety and tolerability of the combination of everolimus and alemtuzumab. (Phase I) II. Determine the maximum tolerated dose of everolimus in this combination. (Phase I) III. Assess the rate of overall responses in patients with relapsed/refractory CLL to treatment with the maximum tolerated dose of everolimus together with a standard dose of alemtuzumab using conventional NCI-WG 1996 response criteria. (Phase II) IV. To assess the complete responses to this combination regimen using conventional NCI-WG 1996 criteria and an expanded definition of response, including CT scans of chest-abdomen-pelvis, immunohistochemical analysis for residual disease in the bone marrow, and sensitive flow cytometry for minimal residual disease in patients in complete clinical remission. V. To monitor and assess toxicity of this regimen. SECONDARY OBJECTIVES: I. To determine the overall and progression-free survival, duration of response, and time to next treatment. II. To assess the correlation between the individual prognostic markers (17p-, p53 gene mutations, 11q-, unmutated VH gene, use of VH3-21, ZAP70+, CD38+, CD49d, B2 microglobulin) and clinical outcome. III. Serial measurement of clinical status and lymphocyte counts to test the rate of reduction in CLL tumor burden. TERTIARY OBJECTIVES: I. Determine the effect of everolimus on the sensitivity of CLL cells to alemtuzumab CDC and ADCC. II. Determine the effect of everolimus on the CLL cell-stroma interaction. III. Detail the in vivo effect of the everolimus-alemtuzumab regimen on critical aspects of the immune system in CLL. OUTLINE: This is a phase I, dose escalation study of everolimus followed by a phase II study. Patients receive oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 7 weeks in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically for up to 5 years. PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
Inclusion

* Diagnosis of CLL manifested by minimum threshold peripheral lymphocyte count of > 5 x 10^9/L (CLL variant) OR palpable adenopathy >= 1cm or clinically palpable splenomegaly (SLL variant); AND immunophenotypic demonstrations of a population of B lymphocytes (as defined by CD19+) which are monoclonal (by light chain exclusion)
* CLL will be diagnosed if these cells have >= 3 of the following characteristics: CD5+, CD23+, dim surface light chain expression, dim surface CD20 expression, AND FISH analysis is negative for IGH/CCND1 and/or immunostaining is negative for cyclin D1 expression to exclude mantle cell lymphoma Previous treatment for CLL Progressive disease: symptomatic CLL (weight loss>10% within 6 months, extreme fatigue, fevers>38.5 C, drenching night sweats without evidence of infection) OR evidence of progressive bone marrow failure (hemoglobin<11g/dL, platelet count<100 x 10^9/L) OR massive (>6 cm below left costal margin) or progressive palpable splenomegaly OR massive (>10 cm) or measurable and progressive lymphadenopathy
* Please contact study investigator and/or consult protocol document for specific details on laboratory criteria CD52 expression by CLL cells Willing to provide mandatory biospecimen samples for research studies as required by the protocol Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only Willingness to return to the enrolling institution for follow-up
* ECOG Performance Status (PS) 0, 1, or 2--Exceptions: Grade 3 allowed if caused by CLL and not other co-morbidities Provide informed written consent Life expectancy >= 3 months

Exclusion

* Any of the following comorbid conditions: NYHA class III-IV heart disease, recent myocardial infarction (< 6 months prior to registration), uncontrolled infection, infection with the human immunodeficiency virus (HIV/AIDS), serological evidence of active hepatitis B infection (HBsAg or HBeAg positive) or positive hepatitis C serology, as further severe immunosuppression with this regimen may occur
* Evidence of active autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia Other active primary malignancy requiring treatment or that limits survival to =< 2 years Any major surgery =< 4 weeks prior to registration Concurrent investigational drug therapy Any of the following: pregnant women,nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, abstinence, etc.)
* Concomitant use of the following CYP3A4 strong inhibitors: Clarithromycin, Nefazodone, Telithromycin, Aprepitant, Indinavir, Nelfinavir, Diltiazem, Borisonazole, Itrazonazole, Ritonavir, Erythromycin, Ketoconazole, Saquinavir, Fluconazole (may be used if drug levels can be monitored)
* Patients with any known bleeding diathesis (any congenital bleeding disorder that affects platelet function and/or coagulation including von Willebrand's Disease)
* Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air Receiving anticoagulant therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Zent, M.D., Study Chair — Mayo Clinic; Jose F. Leis, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Dose Level 1; Phase 2, Dose Level 1: Patients receive 2.5mg of oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 8 weeks.
- Phase 1, Dose Level 2: Patients receive 5mg of oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 8 weeks.
Period: Overall Study
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 2, Dose Level 1
Started | 7 | 9 | 12
Completed | 6 | 6 | 12
Not Completed | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 2, Dose Level 1 | Total
Number analyzed (Participants) | 6 | 6 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 72.5 [66 to 78] | 73 [54 to 82] | 71 [61 to 82] | 72 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 2 | 2 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12 | 24
Previouse number of regimens [Median (Full Range); unit: regimens] | 2 [1 to 6] | 3.5 [1 to 5] | 3 [1 to 10] | 3 [1 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response (Complete or Partial Remission)
Description: CR requires all of the following for a period of at least 2months:Absence of lymphadenopathy.No hepatomegaly or splenomegaly.Absence of constitutional symptoms.• Neutrophils>1500/ul•Platelets>100,000/ul • Hemoglobin >11.0gm/dl• Peripheral blood lymphocytes <4000/uLBonemarrow. normocellular with<30%of nucleated cells being lymphocytes.PR requires two for 2+months.≥50%decrease in peripheral blood lymphocyte count from the pretreatment baseline value.≥ 50%reduction in the sum of the products of the maximal perpendicular diameters of the largest measured node or nodal masses in the right and left cervical, axillary, and inguinal lymph node regions.≥ 50%reduction in size of liver and/or spleen noting the maximal distance below the respective costal margins of palpable hepatosplenomegaly during rest.Neutrophils>1500/ul or50%improvement over baseline. Platelets>100,000/ul or50%increase over baseline. Hemoglobin>11.0 gm/dl or50%increase over baseline without transfusions
Time Frame: After 2 courses of treatment
Population: All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
Measure: Number; unit: participants
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 2, Dose Level 1
Number analyzed (Participants) | 6 | 6 | 12
participants
  Complete Response | 0 | 1 | 0
  Partial Response | 3 | 1 | 3

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: The maximum tolerated dose is the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. Dose-limiting toxicity will be defined as an adverse event attributed (definitely, probably, or possibly) to the study treatment and meeting the following criteria.
  Hematologic: ANC ≤ 0.3 x 109/L or platelet count < 10 x 109/L Other nonhematologic: ≥grade 3 as per NCI Common Terminology Criteria for Adverse Events v3.0 except for fatigue, hyperlipidemia, and hyperglycemia.
Time Frame: 1 Month
Population: All phase 1 patients are evaluable
Measure: Number; unit: participants with DLTs
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2
Number analyzed (Participants) | 6 | 6
participants with DLTs | 1 | 2
Statistical Analysis 1: Comparison: Phase 1, Dose Level 1 vs Phase 1, Dose Level 2; Test type: Other; Estimated maximum tolerated dose was 2.5mg of oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 8 weeks

3. Primary Outcome: Test the Safety and Tolerability of the Combination of Everolimus and Alemtuzumab.
Description: The number and severity of all adverse events will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group. Below is the number of patients that experienced a grade 3+ Adverse event that was at least possibly related to Treatment.
Time Frame: Up to 12 months past final treatment
Measure: Number; unit: participants
Groups:
- All Evaluable Patients: Patients receive oral everolimus thrice weekly for 9 weeks and alemtuzumab subcutaneously thrice weekly for 8 weeks.
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 24
participants | 16

4. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 24
Months | 29.5 [11.9 to 36.8]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival time is defined as the time from registration to progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 24
Months | 4.9 [3.4 to 8.1]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a clinical response as the date at which the patient's objective status is first noted to be a Complete Response or Partial Response to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier
Time Frame: up to 5 years
Population: These are 8 patients with verified complete or partial responses(used in primary outcome measure) as well as 2 non verified partial responses.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Evaluable Patients: Patients are only evaluable for duration of response when they have already been noted as a complete response or partial response.
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 10
Months | 4.6 [.7 to 28.4]

7. Secondary Outcome: Time to Subsequent Therapy
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 24
Months | 13.9 [5.5 to 26.3]

ADVERSE EVENTS:
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 2, Dose Level 1
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/9 | 0/12
Other Adverse Events (participants affected / at risk) | 7/7 | 8/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (N=7) | Phase 1, Dose Level 2 (N=9) | Phase 2, Dose Level 1 (N=12)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (N=7) | Phase 1, Dose Level 2 (N=9) | Phase 2, Dose Level 1 (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (7) | 3 (4) | 1 (2)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 2 (2)
Fever (General disorders) | 4 (8) | 2 (2) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0) | 3 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (2) | 1 (1) | 4 (6)
Pharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (3) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (5) | 2 (3) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 5 (7) | 8 (14) | 11 (28)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (12) | 11 (29)
Neutrophil count decreased (Investigations) | 5 (9) | 5 (9) | 7 (19)
Platelet count decreased (Investigations) | 5 (6) | 5 (6) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 6 (10)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes